CLINICAL TRIAL: NCT00281801
Title: Survival in Allogeneic Bone Marrow Transplantation: The Relative Importance of Inpatient Lay Care-Partner Support
Brief Title: Caregiver Support in the Quality of Life of Patients Who Are Undergoing Donor Bone Marrow Transplantation
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCF6330; P30CA043703 (NIH); CCF-6330 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: psychosocial assessment and care — psychosocial assessment and care
Procedure: Quality of Life Assessments — PACT Scale, Brief COPE, POMS Short Form and FACT BMT

SUMMARY:
RATIONALE: Questionnaires that measure quality-of-life may improve the health care team's ability to plan supportive care for patients undergoing donor bone marrow transplantation.

PURPOSE: This clinical trial is studying quality of life in patients who are undergoing donor bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate the relative importance of having a consistent inpatient lay care-partner for patients undergoing allogeneic bone marrow transplantation.

OUTLINE: Patients complete a 30-minute quality of life questionnaire in order to measure their psychosocial health while in the bone marrow transplant program, including Functional Assessment of Cancer Therapy (FACT), Profile of Mood State (POMS), and Brief COPE questionnaires, at the baseline (pre-transplant) appointment, at the first physician's visit after discharge, at day 100 post-transplant, and then at 6 months and 1 year post-transplant. Caregivers complete a 30-minute coping questionnaire at the pre-transplant appointment, at the first physician's visit after discharge, and then at day 100 post-transplant. Caregivers also keep a weekly log of the time spent with the patient in the hospital.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must be a candidate for allogeneic unrelated or related stem cell transplantation

PATIENT CHARACTERISTICS:

* Both patient and lay care-partner must have the ability to understand and the willingness to sign a written informed consent document

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allogeneic Bone Marrow Transplant patients with lay care-partners.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Correlate presence of a lay care-partner with survival post transplant | At least one year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Brian J. Bolwell, MD, Study Chair — Cleveland Clinic Taussig Cancer Institute
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States